CLINICAL TRIAL: NCT06952686
Title: A Seamless Phase 1/3, Multicenter, Single Dose Systemic Gene Transfer Study to Evaluate the Safety, Tolerability, and Efficacy of SRP-9005 in Limb Girdle Muscular Dystrophy Type 2C/R5 Subjects (COMPASS)
Brief Title: A Study of SRP-9005 in Limb Girdle Muscular Dystrophy Type 2C/R5 Pediatric and Adult Participants
Acronym: COMPASS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was Withdrawn per Sponsor decision.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9005-101
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Muscular Dystrophies, Limb-Girdle
Keywords: SRP-9005; Type 2C/R5; LGMD2C/R5; Pediatric; Non-ambulatory; Ambulatory; Phase 1; Phase 3
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle | interventions — Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Intervention Model Description: This study comprises 2 parts: Part A is the Phase 1 portion, Part B is the Phase 3 expansion portion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP-9005 (Experimental): Participants will receive a single intravenous (IV) infusion of SRP-9005.
  Interventions: Biological: SRP-9005; Drug: Corticosteroid

INTERVENTIONS:
Biological: SRP-9005 — Solution for single IV infusion
  Other Names: rAAVrh74.MHCK7.hSGCG
Drug: Corticosteroid — Oral tablet (prophylactic)
  Other Names: Prednisone or equivalent

SUMMARY:
This is a study of a single systemic dose of SRP-9005 in pediatric and adult participants with limb girdle muscular dystrophy type 2C/R5 (LGMD2C/R5). It is comprised of 2 parts (Part A, Part B) that will assess safety and efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

* Ambulatory, defined as able to walk without assistive aid, 10MWR <30 seconds, and NSAD total score ≥20
* Non-ambulatory, defined as 10MWR ≥30 seconds or unable to perform, and PUL 2.0 entry scale score ≥3
* Possess 1 homozygous or 2 heterozygous pathogenic and/or likely pathogenic gamma-SG deoxyribonucleic acid (DNA) gene mutations as documented prior to pre-Infusion screening. Results to be confirmed by sponsor at a CLIA/CAP/ISO15189 certified laboratory prior to dosing.
* Have AAVrh74 antibody titers <1:400 (that is, not elevated) as determined by an enzyme-linked immunoassay

Key Exclusion Criteria:

* Has a symptomatic infection (for example, upper respiratory tract infection, pneumonia, pyelonephritis, meningitis) within 4 weeks before study treatment infusion
* Part A: Has left ventricular ejection fraction (LVEF) <50% on the screening echocardiogram (ECHO) (without use of cardiac medication) or clinical signs and/or symptoms of cardiomyopathy or any history of cardiac disease
* Part B: Has LVEF <40% on the screening ECHO or clinical signs and/or symptoms of cardiomyopathy
* Has FVC <40% of predicted value at screening and/or requirement for nocturnal ventilation
* Serological evidence of current, chronic, or active human immunodeficiency virus infection, or hepatitis B or C infection or active viral or bacterial infection based on clinical observations
* Any prior treatment with gene therapy, cell-based therapy (for example, stem cell transplantation), clustered regularly interspaced short palindromic repeats/CRISPR-associated protein 9 (CRISPR/Cas9), or any other form of gene editing
* Treatment with human growth factor within 3 months of Day 1
* Treatment with any investigational medication within 6 months of the screening visit
* Is unable to undergo or tolerate a cardiac MRI procedure for any reason

Note: Other inclusion/exclusion criteria may apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2032-03-30 (Estimated)

PRIMARY OUTCOMES:
Part A : Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Baseline through Month 60
Part A and B: Change from Baseline in gamma-Sarcoglycan (SG) Expression at Day 60 Post-dose in Ambulatory Participants as Measured by Immunofluorescence (IF) Percent Positive Fibers (PPF) | Baseline, Day 60

SECONDARY OUTCOMES:
Part A and B: Change from Baseline Through Month 60 in North Star Assessment for Dysferlinopathy (NSAD) Total Score | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Performance of the Upper Limb (PUL) Version 2.0 Total Score | Baseline through Month 60
Part A and B: Change from Baseline through Month 60 in Time to Rise From Floor | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Time to Ascend 4 Steps | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Time to Complete the 10-meter Walk/Run (10MWR) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Time to Complete 100-meter Walk/Run (100MWR) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Timed Up and Go | Baseline through Month 60
Part A and B: Change from Baseline in gamma-SG Expression at Day 60 in Ambulatory Participants Post-dose as Measured by IF Percent Fiber Intensity (PFI) | Baseline, Day 60
Part A and B: Change from Baseline in gamma-SG Expression at Day 60 in Ambulatory Participants Post-dose as Measured by Western Assay | Baseline, Day 60
Part A and B: Change from Baseline to Day 60 in Quantity of gamma-SG Protein Expression in Non-ambulatory Participants as Measured by IF PPF | Baseline to Day 60
Part A and B: Change from Baseline to Day 60 in Quantity of gamma-SG Protein Expression in Non-ambulatory Participants as Measured by IF PFI | Baseline to Day 60
Part A and B: Change from Baseline to Day 60 in Quantity of gamma-SG Protein Expression in Non-ambulatory Participants as Measured by Western Assay | Baseline to Day 60
Part A and B: Change from Baseline to Month 24 in Quantity of gamma-SG Protein Expression as Measured by IF PPF | Baseline to Month 24
Part A and B: Change from Baseline to Month 24 in Quantity of gamma-SG Protein Expression as Measured by IF PFI | Baseline to Month 24
Part A and B: Change from Baseline to Month 24 in Quantity of gamma-SG Protein Expression as Measured by Western Assay | Baseline to Month 24
Part A and B: Change from Baseline Through Month 60 in Creatine Kinase Levels | Baseline through Month 60
Part A and B: Loss of Ambulation | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Skeletal Muscle Magnetic Resonance Imaging (MRI) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Wearable Device Stride Velocity 95th Percentile (SV95C) (Ambulatory Participants Only) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Forced Vital Capacity (FVC) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Forced Vital Capacity Percent Predicted (FVC%p) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Forced Expiratory Volume in 1 Second (FEV1) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Forced Expiratory Volume in 1 Second % Predicted (FEV1%p) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Peak Expiratory Flow Rate (PEFR) | Baseline through Month 60
Part A and B: Change from Baseline through Month 60 in Pulmonary Functions as Assessed by Maximal Inspiratory Pressure (MIP) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Percent Predicted Maximal Inspiratory Pressure (MIP%p) | Baseline through Month 60
Part A and B: Change from Baseline through Month 60 in Pulmonary Functions as Assessed by Maximal Expiratory Pressure (MEP) | Baseline through Month 60
Part A and B: Change from Baseline Through Month 60 in Pulmonary Functions as Assessed by Percent Predicted Maximal Expiratory Pressure (MEP%p) | Baseline through Month 60
Part B: Number of Participants with TEAEs | Baseline through Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States